CLINICAL TRIAL: NCT03464955
Title: Virtual Reality Usage in Non-Invasive Surgical Sub-Specialty Procedures
Brief Title: VR Usage in Non-Invasive Surgical Sub-Specialty Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Samuel Rodriguez, Assistant Professor, Department of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 42351
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Stress, Emotional; Stress, Psychological; Behavioral Symptoms
MeSH Terms: conditions — Stress, Psychological; Behavioral Symptoms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The control group will be provided standard of care, which is no use of technologies.
- Intervention Group with Passive Content (Experimental): Interventional arm will use technology based distractions (VR headsets, AR headset, tablets, or BERT projector) to prevent high anxiety before non-invasive surgical subspecialty procedures.
  Interventions: Behavioral: Technology Based Distractions
- Intervention Group with Active Content (Experimental): Interventional arm will use technology based distractions (VR headsets, AR headset, tablets, or BERT projector) to prevent high anxiety before non-invasive surgical subspecialty procedures.
  Interventions: Behavioral: Technology Based Distractions

INTERVENTIONS:
Behavioral: Technology Based Distractions — Technology based distractions (VR headsets, AR headset, tablets, or BERT projector)
  Arms: Intervention Group with Active Content; Intervention Group with Passive Content

SUMMARY:
Preprocedural, preoperative, and prevascular access anxiety in pediatric patients has been previously shown to increase the likelihood of family stressors, agitation, sleep disturbances, and negative behavioral changes. The purpose of this study is to determine if a non-invasive distracting device (Virtual Reality (VR) headset, Augmented Reality (AR) headset, or bed mounted Video Projection unit (i.e. BERT, Bedside EnterRtainment Theater)) is more effective than the standard of care (i.e., no technology based distraction) for preventing anxiety before non-invasive surgical sub-specialty procedures among children during out-patient clinic visits. Examples of the most common procedures include, but are not limited to gastrostomy tube exchanges, suture removals, dressing changes, foley insertions, EEG set up, chest tube removals, cast removals, pin removals and other similar procedures. (The investigators refer to these procedures under an umbrella term of non-invasive surgical subspecialty procedures). The anticipated primary outcome will be reduction of child's anxiety during and after procedures.

DETAILED DESCRIPTION:
Anxiety among children undergoing non-invasive surgical subspecialty procedures is common. Not only is high anxiety traumatic, but research in a surgical setting indicates that high anxiety in children before surgery leads to adverse outcomes such as increased pain and analgesics requirements, delayed hospital discharge and maladaptive behavioral changes. Treating anxiety may decrease any of these undesirable behaviors that may arise when experiencing a non-invasive surgical subspecialty procedure in a clinical setting.

In this study, investigators hope to determine if technology based distractions (VR headsets with headphones, AR headset, or BERT projector) are more effective than standard care for preventing high anxiety before non-invasive surgical subspecialty procedures. As a secondary objective of the study, the investigators seek to determine if the use of technology based distraction will result in higher parent and patient satisfaction as well as evaluate which techniques are most effective. As a tertiary aim, the investigators seek to understand if passive or active interventions are more effective in decreasing anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. Be between ages of 2-18 years of age
2. Have comprehension of instructions in the English language
3. Have parental consent
4. Pediatric patients must be undergoing non-invasive surgical subspecialty procedures at an Lucile Packard Children's Hospital (LPCH) out-patient clinic
5. Children who are normally healthy (ASA I) or have a mild systemic disease (ASA II,III)

Exclusion Criteria:

1. Significant cognitive impairment/developmental delays per parental report or H&P.
2. Children with ASA IV (severe systemic disease that is a constant threat to life) or ASA V (unstable patients not expected to survive >24 hours or without the operation)
3. Children currently taking psychotropic mediations will be excluded from this study due to the affect emotion modulation
4. Strong parental or patient preference for pharmacological anxiolytic
5. Strong parental or patient preference for specific anxiety-reducing technique

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 291 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-11 (Actual)

PRIMARY OUTCOMES:
Change in Pain Score | Immediately Post Non-Invasive Surgical Subspecialty Procedure Minus Baseline
  Peak Pain Score minus Baseline Pain Score. Pain scores range from 0 to 10. 0 represents no pain and 10 represents the worst pain possible. Change in pain score ranges from +10 to -10. Higher positive values represent a worse outcome, and higher negative values represent a better outcome.

SECONDARY OUTCOMES:
Anxiety Score | Immediately Post Non-Invasive Surgical Subspecialty Procedure Minus Baseline
  Fear Faces. Images of faces depicting increasing levels of fear measure the degree of fear the patient is experiencing. Faces correlate to a score ranging from 0 to 4. 0 represents the least scared and 4 represents the most scared. Higher values represent a worse outcome.
Anxiety Meter | Immediately Post Non-Invasive Surgical Subspecialty Procedure Minus Baseline
  Childhood Anxiety Meter
Family Satisfaction | Immediately Post Non-Invasive Surgical Subspecialty Procedure
  Family Satisfaction Survey
Patient Satisfaction | Immediately Post Non-Invasive Surgical Subspecialty Procedure
  Patient Satisfaction Survey
Patient Cooperation | At the time of Non-Invasive Surgical Subspecialty Procedure
  Brief Behavioral Distress Scale (BBDS). Measures patient cooperation. Behavior cooperation choices exist on a scale consisting of non-interfering behaviors, potentially-interfering behaviors and interfering behaviors. Non-Interfering Behaviors = minor, verbal/vocal distress, moan, comfort seeking, etc. Potentially Interfering Behaviors = intense verbal/vocal distress, scream, shout, tensing of muscles, clench, flinch, gritting of teeth, etc.Interfering Behaviors = escape, disrupt, avoid, aggress, etc. Interfering behaviors represent a worse outcome.
Patient Compliance | At the time of Non-Invasive Surgical Subspecialty Procedure
  Modified Induction Compliance Checklist
Parent Pain Catastrophizing Scale (PCS-P) | Baseline and Immediately Post Non-Invasive Surgical Subspecialty Procedure
  PCS-P. Measures the extent of thought concerning pain Scale ranges from 1 to 5. 1 represents not thinking at all about pain and 5 represents thinking very much about pain. Higher values represent a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodriguez, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No